CLINICAL TRIAL: NCT00068198
Title: Evaluation of Human Immune Response to Smallpox Vaccine (Vaccinia Virus)
Brief Title: Human Immune Responses Smallpox
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02-067
Record Dates: First submitted 2003-09-09; First posted 2003-09-10 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2006-05

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — Smallpox Vaccine

INTERVENTIONS:
Biological: Dryvax

SUMMARY:
The purpose of this study is to attempt to identify the immune response of healthy adults to an investigational dilution of the Dryvax smallpox vaccine. In addition, we will try to determine whether certain genetic characteristics influence the size of the sore around the vaccination site, and use blood samples from subjects in the study to make a new form of antibody that could be given to people with vaccine side effects.

DETAILED DESCRIPTION:
Smallpox is a very serious disease that is fatal in about 1 in 3 patients. Smallpox does not exist naturally in the world, and there have been no cases of smallpox in the world since 1980. Smallpox can be prevented through the use of a very effective vaccine called vaccinia virus (Dryvax). After the world was considered free of smallpox, the production of smallpox vaccine was discontinued, but due to the recent concern that the smallpox virus may be used as a means of bioterrorism, the production of the smallpox vaccine may be restarted. Although Dryvax is known to be an effective vaccine for the prevention of smallpox, very little is known about the ability of the body to develop defenses to prevent disease (immune responses) with this vaccine. As new vaccines for preventing smallpox are developed, it will be important to compare the immune responses they cause to the responses that occur with the standard vaccine, Dryvax.

ELIGIBILITY:
Inclusion Criteria:

* Hematocrit greater than 34% for women, greater than 38% for men, white blood cells between 2500 and 11000/mm3 with normal differential, and platelet count equal to or greater than 150000/mm3
* Availability for followup for the planned duration of the study
* Negative urine or serum pregnancy test on day of vaccination for women
* If the subject is female, she agrees to use acceptable contraception and not become pregnant for at least seven months after vaccination
* Negative ELISA for HIV or negative Western Blot for subject who have a positive ELISA and participated in an HIV vaccine trial
* Meets the criteria for assignment into one of the three study groups
* Willing to sign informed consent
* ALT greater than 1.5 times institutional upper limit of normal
* Negative hepatitis B surface antigen and negative antibody to hepatitis C virus
* Negative urine glucose by dipstick
* Adequate renal function defined as a serum creatinine greater than 1.5 mg/dL, urine protein greater than 100 mg/dL or less than 2+ proteinuria, and a calculated creatinine clearance greater than 55 mL/min
* Acceptable medical history by screening evaluation and brief clinical assessment

Exclusion Criteria:

* History of immunodeficiency
* Known or suspected impairment of immunologic function including but not limited to clinically significant liver disease, diabetes mellitus, moderate to severe kidney impairment
* Malignancy other than squamous cell or basal cell skin cancer
* Autoimmune disease
* Live attenuated vaccines within 60 days of study
* Known allergies to any component of the vaccine (e.g. polymyxin B sulfate, dihydrostreptomycin sulfate, chlortetracycline hydrochloride, neomycin sulfate)
* Known allergies to any known component of VIG i.e. thimerosal or previous allergic reaction to immunoglobulins
* Acute febrile illness on the day of vaccination
* Eczema of any degree or history of eczema
* Use of immunosuppressive medication. Corticosteriod nasal sprays are permissible
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol
* History of "illegal" injection drug use
* Inactivated vaccine 14 days prior to vaccination
* Use of experimental agents within 30 days prior to study
* Receipt of blood products or immunoglobulin in the past 6 months
* Pregnant or lactating women
* History of chronic exfoliative skin disorders/conditions
* Any acute skin disorders of large magnitude e.g. laceration requiring sutures, burn greater than 2 x 2 cm
* Any condition that, in the opinion of the investigator, might interfere with study objectives
* Known allergies to any known component of the diluent (i.e. glycerin and phenol)
* Known allergies to cidofovir or probenecid
* Household contacts/sexual contacts with, or occupational exposure to (other than minimal contact), any of the following: 1) pregnant women, 2) children less than 12 months of age, 3) people with a history of eczema, 4) people with chronic exfoliative skin disorders/conditions or any acute skin disorders of large magnitude e.g. laceration requiring sutures, burn greater than 2 x 2 cm, or 5) people with immunodeficiency disease or use of immunosuppressive medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Study Completion 2004-11

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester School of Medicine, Rochester, New York, United States